CLINICAL TRIAL: NCT05248672
Title: A Phase 1 Study to Assess the Pharmacokinetics of Different Multiple Dose Regimens of CT1812 in Older Healthy Volunteers
Brief Title: Study to Assess the Pharmacokinetics of CT1812 in Older Healthy Volunteers
Acronym: COG0107
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: COG0107
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Open Label Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 150 mg QD (Experimental): CT1812 150 mg QD
  Interventions: Drug: CT1812
- 150 mg BID (Experimental): CT1812 150 mg BID
  Interventions: Drug: CT1812
- 300 mg QD (Experimental): CT1812 300 mg QD
  Interventions: Drug: CT1812

INTERVENTIONS:
Drug: CT1812 — Study Drug

SUMMARY:
This an open label study to assess the pharmacokinetics of CT1812 in normal healthy volunteers.

DETAILED DESCRIPTION:
Open label study to assess PK in 36 older healthy volunteers. Subjects will be screened 35 days prior dose to determine eligibility. On day -1 subjects will be admitted to the clinical research unit and on day 1 will be randomized to receive one of the following doses: 150 mg BID, 150 mg QD or 300 mg QD in the fed state. Subjects will be confined in the Clinical Research Unit where they will continue to receive study drug and complete safety assessments, PK and CSF draws, until day 16 when they will be discharged.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women 50-80 years of age, inclusively
* In good health as determined by the Investigator with no clinically significant abnormalities
* Weight between 50.0 and 100.0 kg, inclusive at Screening
* No suicidal ideation
* No active depression
* Living independently at home or in a community setting
* Able to swallow CT1812 capsule or capsules
* Non-smoker with no history of using tobacco or any nicotine-containing products
* Subjects with negative serology for HIV, Hepatitis B, and C
* Negative results for drugs of abuse, cotinine, and alcohol
* Negative test results for COVID-19
* Willing to comply with Clinical Pharmacology Unit's COVID-19 policies

Exclusion Criteria:

* Any chronic medical condition which, in the opinion of the investigator, might pose a safety risk to the subject or interfere with study interpretation
* Subject with active or recent infection requiring antibiotic therapy
* Medical history of vasculitis or any autoimmune disease
* Any recent hospitalization
* Subjects living in a continuous care nursing facility
* Any contraindication to a lumbar puncture
* Subjects with self-reported history of major depression
* History of diabetes
* Intake of drugs or substances potentially involved in clinically significant induction or inhibition of CYP3A4 or P-gp mediated drug interactions with CT1812
* Intake of investigational drug prior to study drug administration on Day 1
* Participation in an investigational device study prior to study drug administration on Day 1
* Grapefruit, grapefruit juice, and Seville oranges/juice must be avoided within 14 days prior to dosing and throughout the course of the study
* Suspected or known drug or alcohol abuse,
* Excessive consumption of coffee, tea, cola, or other caffeinated beverages
* Loss or donation of blood; nation of bone marrow or peripheral stem cells; or donation of plasma
* Venous access considered inadequate; history or evidence of adverse symptoms associated with phlebotomy or blood donation
* Suspected or known allergy to any component of the study treatments
* Employee or family member of the Investigator, study site personnel, or Sponsor
* A subject with any condition that, in the opinion of the Investigator, makes the subject unsuitable for study participation will be excluded

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) in plasma | Day 13 and 15.
  Cmax: Maximum observed plasma concentration occurring at Tmax
Pharmacokinetics (PK) in plasma | Day 13 and 15.
  Tmax: The first time to maximum observed concentration sampled during a dosing interval.
Pharmacokinetics (PK) in plasma | Day 13 and 15.
  Ctau: Concentration at the end of the dosing interval (12 hr for BID group; 24 hr for QD group).
Pharmacokinetics (PK) in plasma | Day 13 and 15.
  AUC 0-12h: Area under the concentration-time curve (AUC) from time 0 to 12 hours post-dose.
Pharmacokinetics (PK) in plasma | Day 13 and 15.
  AUC 0-24h: AUC from time 0 to 24 hours post-dose.
Pharmacokinetics (PK) in plasma | Day 13 and 15.
  AUC 0-last: AUC from time 0 to the time of the last measurable concentration at 48 and 72 hours as applicable.
Pharmacokinetics (PK) in plasma | Day 13 and 15.
  AUC 0-inf: Area under the concentration-time curve (AUC) from time 0 extrapolated to infinity, calculated using the observed value of the last non-zero concentration.
Pharmacokinetics (PK) in plasma | Day 13 and 15.
  AUC_%Extrap: Percent of AUC0-inf contributed by extrapolation beyond AUC0-last.
Pharmacokinetics (PK) in plasma | Day 13 and 15.
  λz : Terminal elimination phase rate constant.
Pharmacokinetics (PK) in plasma | Day 13 and 15.
  t½: Terminal phase half-life.
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  Cmax - Maximum observed plasma concentration occurring at Tmax.
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  Tmax -The first time to maximum observed concentration sampled during a dosing interval.
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  Cavg,ss - Average plasma concentration at steady-state interval.
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  Ctau-Concentration at the end of the dosing interval (12 hr for BID group; 24 hr for QD group).
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  Fluctuation (%) - Fluctuation (%) between maximum and minimum concentrations over the steady-state dosing interval.
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  AUC-0-tau - Area under the concentration-time curve from time 0 to the end of the dosing interval (0-12 for the BID group; 0 - 24 for the QD groups) .
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  λz- Terminal elimination phase rate constant
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  t½ - Terminal phase half-life
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  AUCcum- Accumulation ratio in AUC, calculated as AUC0-tau,ss/AUC0-tau,D1
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  Ctau,cum- Accumulation ratio in Ctau, calculated as Ctau,ss/Ctau,D1
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF). | Day 13 and 15.
  Cmax,cum - Accumulation ratio in Cmax, calculated as Cmax,ss/Cmax,D1
Pharmacokinetics (PK) in Cerebrospinal Fluid (CSF)- CSF/plasma ratio | Day 13 and 15.
  CSF/plasma ratio - Pre-dose on Day 13 and 3h (±15 min) post-dose on Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Caggiano, MD, Study Director — Cognition Therapeutics
Locations (1):
- Accel Clinical Research, DeLand, Florida, United States

IPD SHARING:
Plan to Share IPD: No